CLINICAL TRIAL: NCT04167345
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of VX-814 in PiZZ Subjects
Brief Title: Evaluation of the Efficacy and Safety of VX-814 in Subjects With the PiZZ Genotype
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: at Sponsor's discretion
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX19-814-101
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Parts A1, A2 and B Combined: Placebo (Placebo Comparator): Participants received placebo matched to VX-814 in the treatment period for 28 days.
  Interventions: Drug: Placebo
- Part A1: VX-814 100 milligrams (mg) (Experimental): Participants received VX-814 100 mg every 12 hours (q12h) in the treatment period for 28 days.
  Interventions: Drug: VX-814
- Part A1: VX-814 200 mg (Experimental): Participants received VX-814 200 mg q12h in the treatment period for 28 days.
  Interventions: Drug: VX-814
- Parts A1 and A2 Combined: VX-814 400 mg (Experimental): Participants received VX-814 400 mg q12h in the treatment period for 28 days.
  Interventions: Drug: VX-814
- Part B: VX-814 600 mg (Experimental): Participants received VX-814 600 mg q12h in the treatment period for 28 days.
  Interventions: Drug: VX-814

INTERVENTIONS:
Drug: VX-814 — Tablet for oral administration.
  Arms: Part A1: VX-814 100 milligrams (mg); Part A1: VX-814 200 mg; Part B: VX-814 600 mg; Parts A1 and A2 Combined: VX-814 400 mg
Drug: Placebo — Placebo matched to VX-814 for oral administration.
  Arms: Parts A1, A2 and B Combined: Placebo

SUMMARY:
This study will evaluate the efficacy, safety and pharmacokinetics (PK) of VX-814 in PiZZ subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects must have a PiZZ genotype confirmed at screening
* Plasma AAT levels indicating severe deficiency at screening

Key Exclusion Criteria:

* History of a medical condition that could negatively impact the ability to complete the study
* Solid organ, or hematological transplantation or is currently on a transplant list
* History of use of gene therapy or RNAi therapy at any time previously

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Davis Medical Center, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Shands Hospital, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Blessing Corporate Services, Inc., dba Blessing Health System, Hannibal, Missouri
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Renovatio Clinical, Houston, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- Canada (2):
  - Queen Elizabeth II Health Sciences Center, Halifax
  - Inspiration Research Ltd, Toronto
- Germany (3):
  - University Hospital RWTH Aachen, Aachen
  - Universitätsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
- Royal College of Surgeons in Ireland Clinical Research Centre, Beaumont Hospital, Beaumont, Ireland

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 3 parts in the study: Parts A1, A2 and B. As pre-specified in SAP, data collected for the placebo group for Parts A1, A2 and B were pooled and reported as a single combined arm (Parts A1, A2 and B Combined: Placebo) and data collected for VX-814 400 mg for Parts A1 and A2 were pooled and reported as a single combined arm (Parts A1 and A2 Combined: VX-814 400 milligrams [mg]) in the below presented results.
Pre-assignment Details: This study was conducted in participants 18 through 80 of years of age, inclusive with the PiZZ genotype.
Groups:
- Part A1: VX-814 100 mg: Participants received VX-814 100 mg once every 12 hours (q12h) in the treatment period for 28 days.
Period: Overall Study
Arm/Group | Parts A1, A2 and B Combined: Placebo | Part A1: VX-814 100 mg | Part A1: VX-814 200 mg | Parts A1 and A2 Combined: VX-814 400 mg | Part B: VX-814 600 mg
Started | 10 | 4 | 3 | 13 | 18
Completed | 9 | 3 | 3 | 13 | 18
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A1: VX-814 100 mg: Participants received VX-814 100 mg q12h in the treatment period for 28 days.
- Total: Total of all reporting groups
Arm/Group | Parts A1, A2 and B Combined: Placebo | Part A1: VX-814 100 mg | Part A1: VX-814 200 mg | Parts A1 and A2 Combined: VX-814 400 mg | Part B: VX-814 600 mg | Total
Number analyzed (Participants) | 10 | 4 | 3 | 13 | 18 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.3) | 51.8 (14.8) | 55.5 (7.8) | 57.9 (13.2) | 57.9 (9.1) | 56.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 0 | 7 | 12 | 27
  Male | 5 | 1 | 3 | 6 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 9 | 3 | 3 | 12 | 14 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 10 | 4 | 3 | 13 | 18 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Plasma Functional Alpha-1 Antitrypsin (AAT) Levels [Mean (Standard Deviation); unit: micromole per liter] | 4.2 (1.2) | 5.1 (2.3) | 3.9 (0.4) | 3.9 (0.7) | 4.5 (1.0) | 4.3 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Functional Alpha-1 Antitrypsin (AAT) Levels
Time Frame: From Baseline at Day 28
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug. The "overall number of participants analyzed" signifies participants who were evaluable at the specified time point. As pre-specified in SAP, statistical comparison with placebo were planned only for VX-814 400 mg and 600 mg treatment arms.
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Parts A1, A2 and B Combined: Placebo | Part A1: VX-814 100 mg | Part A1: VX-814 200 mg | Parts A1 and A2 Combined: VX-814 400 mg | Part B: VX-814 600 mg
Number analyzed (Participants) | 6 | 2 | 3 | 8 | 15
micromole per liter | -0.4 (0.3) | 0.2 (0.1) | 0.3 (0.5) | 1.4 (0.6) | 1.6 (1.0)
Statistical Analysis 1: Comparison: Parts A1, A2 and B Combined: Placebo vs Parts A1 and A2 Combined: VX-814 400 mg; Test type: Superiority; p < .0001, t-test, 2 sided; Mean Difference = 1.7, 95% CI 2-sided [1.1 to 2.3]
Statistical Analysis 2: Comparison: Parts A1, A2 and B Combined: Placebo vs Part B: VX-814 600 mg; Test type: Superiority; p < .0001, t-test, 2 sided; Mean Difference = 2.0, 95% CI 2-sided [1.1 to 2.9]

2. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 8
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Parts A1, A2 and B Combined: Placebo | Part A1: VX-814 100 mg | Part A1: VX-814 200 mg | Parts A1 and A2 Combined: VX-814 400 mg | Part B: VX-814 600 mg
Number analyzed (Participants) | 10 | 4 | 3 | 13 | 18
participants
  Participants With AEs | 4 | 3 | 1 | 10 | 14
  Participants With SAEs | 0 | 2 | 1 | 1 | 0

3. Secondary Outcome: Change in Plasma Antigenic AAT Levels
Time Frame: From Baseline at Day 28
Population: FAS. The "overall number of participants analyzed" signifies participants who were evaluable at the specified time point. As pre-specified in SAP, statistical comparisons with placebo were planned only for VX-814 400 mg and 600 mg treatment arms.
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Parts A1, A2 and B Combined: Placebo | Part A1: VX-814 100 mg | Part A1: VX-814 200 mg | Parts A1 and A2 Combined: VX-814 400 mg | Part B: VX-814 600 mg
Number analyzed (Participants) | 6 | 2 | 3 | 8 | 15
micromole per liter | 0.4 (1.3) | 0.1 (0.2) | 0.7 (0.7) | 2.4 (1.2) | 2.6 (1.1)
Statistical Analysis 1: Comparison: Parts A1, A2 and B Combined: Placebo vs Parts A1 and A2 Combined: VX-814 400 mg; Test type: Superiority; p = 0.0114, t-test, 2 sided; Mean Difference = 2.0, 95% CI 2-sided [0.5 to 3.4]
Statistical Analysis 2: Comparison: Parts A1, A2 and B Combined: Placebo vs Part B: VX-814 600 mg; Test type: Superiority; p = 0.0009, t-test, 2 sided; Mean Difference = 2.3, 95% CI 2-sided [1.1 to 3.5]

4. Secondary Outcome: Observed Pre-dose Plasma Concentration of VX-814
Time Frame: Pre-dose at Day 7, Day 14, Day 21, and Day 28
Population: Pharmacokinetic analysis included all randomized participants who received at least 1 dose of study drug. Here "number analyzed" signifies participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Part A1: VX-814 100 mg | Part A1: VX-814 200 mg | Parts A1 and A2 Combined: VX-814 400 mg | Part B: VX-814 600 mg
Number analyzed (Participants) | 4 | 3 | 13 | 18
microgram per milliliter
  Day 7: number analyzed (Participants) | 2 | 3 | 9 | 14
  Day 7 | 0.476 (0.375) | 0.948 (0.512) | 3.53 (1.72) | 10.3 (6.55)
  Day 14: number analyzed (Participants) | 2 | 3 | 8 | 17
  Day 14 | 0.244 (0.0919) | 1.07 (0.152) | 3.25 (2.23) | 8.53 (11.8)
  Day 21: number analyzed (Participants) | 1 | 1 | 6 | 16
  Day 21 | 0.700 | 1.45 | 3.68 (3.40) | 7.20 (6.05)
  Day 28: number analyzed (Participants) | 3 | 3 | 7 | 15
  Day 28 | 0.326 (0.0282) | 0.993 (0.0300) | 3.23 (2.82) | 5.80 (3.73)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 8
Arm/Group | Parts A1, A2 and B Combined: Placebo | Part A1: VX-814 100 mg | Part A1: VX-814 200 mg | Parts A1 and A2 Combined: VX-814 400 mg | Part B: VX-814 600 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4 | 0/3 | 0/13 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/4 | 1/3 | 1/13 | 0/18
Other Adverse Events (participants affected / at risk) | 4/10 | 1/4 | 0/3 | 9/13 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parts A1, A2 and B Combined: Placebo (N=10) | Part A1: VX-814 100 mg (N=4) | Part A1: VX-814 200 mg (N=3) | Parts A1 and A2 Combined: VX-814 400 mg (N=13) | Part B: VX-814 600 mg (N=18)
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Parts A1, A2 and B Combined: Placebo (N=10) | Part A1: VX-814 100 mg (N=4) | Part A1: VX-814 200 mg (N=3) | Parts A1 and A2 Combined: VX-814 400 mg (N=13) | Part B: VX-814 600 mg (N=18)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 6
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 2
Crystal urine present (Investigations) | 0 | 0 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
During the study, elevated liver enzymes (AST/ALT) were observed in several participants and analysis of available pharmacokinetics data indicated that VX-814 exposures achieved were low. Based on these data, Vertex concluded that it would not be feasible to safely reach targeted exposure levels with VX-814. Thus, the study was terminated early at the sponsor's discretion. Given the study was terminated early, the data are incomplete, and results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT04167345/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04167345/SAP_001.pdf